CLINICAL TRIAL: NCT02247180
Title: Cognitive Rehabilitation in Alzheimer's Disease (AD)
Brief Title: Cognitive Rehabilitation in Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Collaborators: German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Principal Investigator, Elisabeth Kasper, Dipl. psych, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A 2014-0113
Record Dates: First submitted 2014-09-16; First posted 2014-09-23 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Rehabilitation (Experimental): cognitive rehabilitation for 12 weeks
  Interventions: Behavioral: cognitive rehabilitation
- Cognitive Training (Active Comparator): standardized cognitive training in the domesticity
  Interventions: Behavioral: standardized cognitive training

INTERVENTIONS:
Behavioral: cognitive rehabilitation
  Arms: Cognitive Rehabilitation
Behavioral: standardized cognitive training
  Arms: Cognitive Training

SUMMARY:
This study aims to proof the efficacy of a cognitive rehabilitation program for patients with mild dementia in Alzheimers Disease with respect to activities of daily living.

DETAILED DESCRIPTION:
This prospective randomized, single blind intervention study aims to proof a cognitive rehabilitation program for patients with mild dementia in Alzheimers Disease (AD). The investigators modified a manualized and established German behavioural therapy program (KORDIAL) to use in a group context. The respective modules contain multimodal and multiprofessional approaches to improve capabilities relevant to activities of daily living (external memory support, compensation strategies, training of everyday competence, communication training). The intervention group receives this therapy for 12 weeks. Age and gender matched participants with AD serve as active control sample receiving a standardized cognitive training in the domesticity. The primary outcome are measurements of skills in activities of daily living prior the intervention as well as at the end of the intervention (after 3 months) and after 6 months (Follow up).

ELIGIBILITY:
Inclusion Criteria:

* mild dementia in Alzheimer's disease (NINCDS-ADRDA)
* Mini Mental State ≥ 17

Exclusion Criteria:

* severe psychiatric disorder
* severe brain disorder (epilepsy, tumor, stroke)
* contraindication for MRI examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in activities of daily living measured by a test for action regulation and planning skills (HOTAP) to the end of intervention and to follow-up (6 months later) | prior intervention, after intervention (3 months), after 6 months
Change from baseline in activities of daily living measured by an ADL-scale (Bayer-ADL) to the end of intervention and to follow-up (6 months later) | prior intervention, after intervention (3 months), after 6 months
Change from baseline in behavioural memory abilities measured by a behavioural memory test (RBMT) to the end of intervention and to follow-up (6 months later) | prior intervention, after intervention (3 months), after 6 months

SECONDARY OUTCOMES:
Change from baseline in general cognitive state measured by the Consortium to Establish a Registry for Alzheimer´s Disease (CERAD) to the end of intervention and to follow-up (6 months later) | prior intervention, after intervention (3 months), after 6 months
Change from baseline in structural and functional connectivity of the brain measured by MRI to the end of intervention and to follow-up (6 months later) | prior intervention, after intervention (3 months), after 6 months
Change from baseline in depression and quality of life measured by two scales (GDS, DEMQoL) to the end of intervention and to follow-up (6 months later) | prior intervention, after intervention (3 months), after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Teipel, Prof., Principal Investigator — Department of Psychosomatic Medicine, University of Rostock, Rostock, Germany
Locations (1):
- Department of Psychosomatic Medicine, University of Rostock, Rostock, Germany